CLINICAL TRIAL: NCT03306407
Title: A Multicentre Intervention Study on the Use of Hand Sanitizers in the Prevention of Intestinal Colonization With Extended-spectrum Beta-lactamase-producing Enterobacteriaceae in Travellers to the Indian Subcontinent
Brief Title: The Effect of Hand Hygiene on Colonization Rates With Multidrug Resistant Enteric Pathogens in Travellers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Hatz (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Christoph Hatz, Prof. Dr. med. Christoph Hatz, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LEK EKNZ 2015-271
Record Dates: First submitted 2015-12-09; First posted 2017-10-11 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Drug Resistance, Multiple; Travel Medicine

ARMS (2):
- Baseline Group (No Intervention): Group screened for colonization with ESBL-producing Enterobacteriaceae pre- and post-travel after having received standard pre-travel advice
- Intervention Group (Active Comparator): Group screened for colonization with ESBL-producing Enterobacteriaceae pre- and post-travel after having received pre-travel advice with special focus on improved hand hygiene including the use of hand gel sanitizer (Hartmann Sterillium) (bundle intervention)
  Interventions: Other: Improved hand hygiene

INTERVENTIONS:
Other: Improved hand hygiene — The intervention group receives pre-travel advice with a special focus on improved hand hygiene including the use of hand gel sanitizer (Hartmann Sterillium) (bundle intervention)
  Arms: Intervention Group

SUMMARY:
Travelling to tropical and subtropical countries is a known risk factor for becoming colonized with extended-spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae. Especially travellers returning from the Indian subcontinent show high colonization rates of up to almost 90%.

While risk factors for becoming colonized have been identified in several studies, no preventive measure has been tested so far.

One of the factors associated with becoming colonized while travelling is suffering from travellers' diarrhoea. Earlier studies looking at diarrhoea in childhood as well as school and/or work absenteeism because of diarrhoeal diseases have shown protective effects through good hand hygiene. Furthermore, a recent retrospective study has shown lower rates of travellers' diarrhoea in people using hand gel sanitizers. Improving hand hygiene in travellers through increased hand washing and the use of hand gel sanitizers might therefore not only decrease the rate of travellers' diarrhoea but the carriage rate with ESBL-producing Enterobacteriaceae as well. However, there is no prospective data available to prove the usefulness of such an intervention, neither in the prevention of travellers' diarrhoea nor in the prevention of colonization.

In the current study, investigators plan to compare colonization rates with ESBL-producing Enterobacteriaceae in travellers receiving pre-travel advice on improved hand hygiene (including the use of hand gel sanitizers) with travelers receiving standard advice.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* travelling to the Indian subcontinent (India, Bhutan and/or Nepal) for up to 4 weeks

Exclusion Criteria:

* age < 18 years
* travelling to other destinations than India, Bhutan and/or Nepal
* antibiotic treatment at the time of the first sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2015-12; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Colonization rates with ESBL-producing Enterobacteriaceae in travellers returning from South Asia | up to 1 week after travel
  Coloinzation rates with ESBL-producing Enterobacteriaceae in travellers

SECONDARY OUTCOMES:
Incidence of travellers' diarrhoea (during and up to 2 weeks after travelling, assessed through self-reporting) | up to 2 weeks after travel
  Incidence of travellers' diarrhoe

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Swiss Tropical and Public Health Institute, Basel
  - Epidemiology, Biostatistics and Prevention Institute, Zurich

REFERENCES:
- [Background] Kuenzli E, Jaeger VK, Frei R, Neumayr A, DeCrom S, Haller S, Blum J, Widmer AF, Furrer H, Battegay M, Endimiani A, Hatz C. High colonization rates of extended-spectrum beta-lactamase (ESBL)-producing Escherichia coli in Swiss travellers to South Asia- a prospective observational multicentre cohort study looking at epidemiology, microbiology and risk factors. BMC Infect Dis. 2014 Oct 1;14:528. doi: 10.1186/1471-2334-14-528. PMID 25270732
- [Background] Kantele A, Laaveri T, Mero S, Vilkman K, Pakkanen SH, Ollgren J, Antikainen J, Kirveskari J. Antimicrobials increase travelers' risk of colonization by extended-spectrum betalactamase-producing Enterobacteriaceae. Clin Infect Dis. 2015 Mar 15;60(6):837-46. doi: 10.1093/cid/ciu957. Epub 2015 Jan 21. PMID 25613287
- [Background] Paltansing S, Vlot JA, Kraakman ME, Mesman R, Bruijning ML, Bernards AT, Visser LG, Veldkamp KE. Extended-spectrum beta-lactamase-producing enterobacteriaceae among travelers from the Netherlands. Emerg Infect Dis. 2013 Aug;19(8):1206-13. doi: 10.3201/eid.1908.130257. PMID 23885972
- [Background] Henriey D, Delmont J, Gautret P. Does the use of alcohol-based hand gel sanitizer reduce travellers' diarrhea and gastrointestinal upset?: A preliminary survey. Travel Med Infect Dis. 2014 Sep-Oct;12(5):494-8. doi: 10.1016/j.tmaid.2014.07.002. Epub 2014 Jul 11. PMID 25065273